CLINICAL TRIAL: NCT00162149
Title: Open-Label, Multiple-Dose, Drug Interaction Study to Assess the Effect of Nevirapine on the Pharmacokinetics of Atazanavir in HIV-Infected Individuals
Brief Title: ATV/Ritonavir Nevirapine Interaction (USPAC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI424-137
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Atazanavir Sulfate; Ritonavir; atazanavir, ritonavir drug combination

ARMS (4):
- A1 (No Intervention)
  Interventions: Drug: Nevirapine
- A2 (Experimental)
  Interventions: Drug: Nevirapine + Atazanavir/Ritonavir
- A3 (Experimental)
  Interventions: Drug: Nevirapine + Atazanavir/Ritonavir
- B1 (No Intervention)
  Interventions: Drug: Atazanavir + Ritonavir

INTERVENTIONS:
Drug: Nevirapine — Tablets, Oral, 200 mg, Twice daily, 3 days.
  Arms: A1
Drug: Nevirapine + Atazanavir/Ritonavir — Tablets + Capsules/Capsules, Oral, 200 mg + 300/100 mg, twice daily + once daily, 10 days.
  Other Names: Reyataz
  Arms: A2
Drug: Nevirapine + Atazanavir/Ritonavir — Tablets + Capsules/Capsules, Oral, 200 mg + 400/100 mg, twice daily + once daily, 10 days.
  Other Names: Reyataz
  Arms: A3
Drug: Atazanavir + Ritonavir — Capsules/capsules, Oral, 300/100 mg, once daily, 10 days.
  Other Names: Reyataz
  Arms: B1

SUMMARY:
Open-Label, multiple-dose, drug interaction study to assess the effect of nevirapine on the pharmacokinetics of atazanavir in HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form
* For Cohort 1, HIV-infected subjects receiving nevirapine 200 mg twice-daily and 2 to 3 NRTIs for at least 6 weeks
* For Cohort 2, HIV-infected subjects receiving atazanavir 300 mg and ritonavir 100 mg once-daily and 2 to 3 NRTIs for at least 6 weeks
* Have had 2 measurements of plasma HIV RNA of <400 copies/mL. The first test being 6 to 16 weeks prior and the second being within 3 weeks prior to Day 1
* Have CD4 cell count >=200 cells/mm3
* Body Mass Index of 18 to 35 kg/m2.
* Men and women, ages 18 to 55.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Presence of a newly diagnosed HIV-related opportunistic infection or CD4 cell count <200 cell/mm3 within the previous 6 months.
* Any significant acute or chronic medical illness, unless stable or controlled by a non-prohibited medication.
* History of virologic failure on an antiretroviral regimen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Steady state pharmacokinetics of atazanavir/ritonavir 300/100mg & 400/100mg each co-administered w/ nevirapine 200mg twice-daily w/ 2 to 3 nucleoside reverse transcriptase inhibitors relative to that of a second cohort of subj.

SECONDARY OUTCOMES:
Steady state PK of 2 atazanavir/ritonavir&nevirapine regimens relative to historic data of atazanavir 400mg in HIV-inf subj;Safety & tolerability of co-admin of atazanavir,ritonavir,&nevirapine in the presence of 2to3 nucleoside rev. transcriptase inhibi

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (2):
  - Local Institution, Pomona, California
  - Local Institution, Seattle, Washington
- Local Institution, London, Greater London, United Kingdom